CLINICAL TRIAL: NCT06091618
Title: Laser Vaporization of the Prostate: Comparative Study Between Ejaculatory Preserving and Non-ejaculatory Preserving Technique
Brief Title: Laser Vaporization of the Prostate: Comparing Between Ejaculatory Preserving and Non-ejaculatory Preserving Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ejaculatory sparing laser turp
Record Dates: First submitted 2023-09-26; First posted 2023-10-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-09

CONDITIONS: Prostatic Hyperplasia
Keywords: ejaculatory preserving; laser vaporization of the prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: prospective, randomized clinical study.
  Exclusion criteria
  * Major psychiatric and somatic diseases and the use of drugs that affect sexual function
  * Patients with ejaculatory dysfunction or no ejaculation
  * Patients with documented or suspected prostate cancer
  * Patients with neurogenic bladder, voiding dysfunction, urethral strictures, and malignancies of the upper or lower urinary tract,
  * Prostates sized more than 80 CC, severe comorbidities or high surgical risk patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new technique of ejaculatory preserving laser vaporization prostatectomy (Active Comparator): laser will be employed to preform vaporization. The ejaculatory preserving procedure will be done in the following steps:
  1. Setting a mark cut 1 cm proximal of the verumontanum as orientation.
  2. Complete resection of the middle lobe to the abovementioned mark.
  3. Vaporization of lateral lobes to the capsule and the ventral side to the level of the verumontanum with avoidance of paracollicular digging.
  4. Circular resection of the internal bladder neck.
  5. Apical resection utilizing the colliculus seminalis as a distal resection border and maintaining a 1cm safety area for preservation of ejaculation.
  6. Total removal of prostate cuts and final check to confirm that there are no obstructive components.
  Interventions: Procedure: new technique of ejaculatory preserving laser prostatectomy
- conventional technique laser vaporization prostatectomy (Active Comparator): non ejaculatory preserving laser vaporization of the prostate
  Interventions: Procedure: conventional technique of laser vaporization of the prostate

INTERVENTIONS:
Procedure: new technique of ejaculatory preserving laser prostatectomy — laser will be employed to preform vaporization. The ejaculatory preserving procedure will be done in the following steps:
  Setting a mark cut 1 cm proximal of the verumontanum as orientation. Complete resection of the middle lobe to the abovementioned mark. Vaporization of lateral lobes to the capsule and the ventral side to the level of the verumontanum with avoidance of paracollicular digging.
  Circular resection of the internal bladder neck. Apical resection utilizing the colliculus seminalis as a distal resection border and maintaining a 1cm safety area for preservation of ejaculation.
  Total removal of prostate cuts and final check to confirm that there are no obstructive components.
  Arms: new technique of ejaculatory preserving laser vaporization prostatectomy
Procedure: conventional technique of laser vaporization of the prostate — conventional laser vaporization of the prostate
  Arms: conventional technique laser vaporization prostatectomy

SUMMARY:
The present work aimed to compare between The Outcomes of conventional technique of laser prostatectomy versus the new ejaculatory sparing technique .

DETAILED DESCRIPTION:
Benign prostate hyperplasia (BPH) is a histological diagnosis which is identified by non-malignant hyperplasia of prostatic tissue due to smooth muscle and epithelial cell proliferation in the prostate transition zone.

The prevalence of histologically diagnosed (BPH) increases from 8% in men aged 31 to 40 years old to 40-50% in men aged 51 to 60 years old. This increases to over 80% in men older than 80 years old.

Bladder outlet obstructions (BOO) are one of the major disorders in the aging male, The most common aetiology of BOO in elderly men above the age of 60 years is (BPH), but younger men (< 50 years old) can also experience infra vesical obstruction from a small but obstructive prostate.

Ejaculation is one of the fundamental domains of male sexual function An almost inevitable adverse event of the conventional TURP is the loss of antegrade ejaculation, seen in 65%-80% of patients.

The use of alpha receptor antagonists is also known to cause a loss in antegrade ejaculation. Aside from peri- and postoperative morbidities, such as bleeding and TURP syndrome, the loss of ejaculation represents a major reason for the avoidance of surgical treatment. This is a particular issue among young people who hesitate to agree to the TURP procedure due to the fear of loss of ejaculation. Losing the ability to ejaculate often leads to a subsequent decrease in sexual pleasure, which has psychosocial implications but can also impact on aspects related to their cultural background, desire for children, and sexual life.

According to the current theory of ejaculation, the loss of antegrade ejaculation is attributed to the loss of bladder neck function after resection.

Even though TURP has a high success rate, the perioperative morbidity and operative safety specially in relation to bleeding pose serious concerns In addition to bleeding, retrograde ejaculation and TURP syndrome due to irrigant absorption are also relevant to intra and postoperative complications.

Despite technical advancements in TURP, blood transfusion rates are still 2 % to 7 %, TUR syndrome occurs in 2 %, stress urinary incontinence in 2 %, retrograde ejaculation in 65 % to 70.0%, urethral strictures in 4 %, bladder neck contractures in 4 % and early revision rates are 3 % to 5 %. These, along with prolonged catheterization time, advocate for alternatives to this treatment modality that offer similar clinical results but fewer complications

Laser vaporization of prostate is one of these methods. Lasers generate different effects in tissues, like coagulation and vaporization. Different types of laser like potassium-titanyl phosphate (KTP), holmium, diode and thulium are available. Of these, those gaining more popularity are the photoselective vaporization of the prostate (PVP) using the KTP laser, and holmium laser enucleation of the prostate (HOLEP).

The semiconductor diode laser is thought to be the best in relation to its haemostatic properties, but due to postoperative dysuria, pain, and storage urinary symptoms, it was less acceptable , A newly introduced diode laser, operating on the wavelength of 980 nm, is different in terms of its new fiber design, greater ablative properties of tissues, and efficient haemostasis due to its significant simultaneous absorption in water and Haemoglobin

The conventional technique of laser prostatectomy is traditionally performed with careful vaporization of apical tissue around the verumontanum.

To preserve the antegrade ejaculation, the paracollicular and the situated tissue, which is located 1 cm proximal to the verumontanum should not be vaporized. This is mainly related to the importance of the musculus ejaculatorius and verumontanum for ejaculation.

Based on this clearer understanding of the process of ejaculation, a new technique of trans urethral laser vaporization of the prostate , termed ejaculation-preserving technique was developed with the overarching aim of preserving antegrade ejaculation with comparable functional outcome for micturition parameters to regular technique.

ELIGIBILITY:
Inclusion criteria:

* Age >45 years old, clinical diagnosis of BOO by medical history and physical examination (including digital rectal examination)
* International prostate symptoms score (IPSS) >14 points
* Normal PSA (PSA<4 ng / ml or free/ total PSA >0.25)
* Prostate size < 80 gm
* Men with recurrent urinary retention (drug-refractory), urinary infection, or haematuria who had failed standard medical therapy (alpha-blockers, 5-alpha reductive inhibitors)
* Patients were also required to have an active and healthy sexual life, the ability to ejaculate and a desire to preserve ejaculation

Exclusion criteria

* Major psychiatric and somatic diseases and the use of drugs that affect sexual function
* Patients with ejaculatory dysfunction or no ejaculation
* Patients with documented or suspected prostate cancer
* Patients with neurogenic bladder, voiding dysfunction, urethral strictures, and malignancies of the upper or lower urinary tract,
* Prostates sized more than 80 CC, severe comorbidities or high surgical risk patients.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-27 (Estimated); Study Completion 2024-04-27 (Estimated)

PRIMARY OUTCOMES:
compare between The Outcomes of conventional technique of laser prostatectomy versus the new ejaculatory sparing technique regarding semen volume | one year
  decreased,vanished or the same
maximum flow rate of the urine after the procedure (Qmax ) | one year
  maximum flow rate increased or decreased or the same Qmax Interpretation * is higher than 15ml/sec Normal 10-15ml/sec Equivocal is lower than 10ml/sec Obstruction or weak detrusor
international prostate symptoms score (IPSS) | one year
  Score: 1-7: Mild 8-19: Moderate 20-35: Severe
  1. Incomplete Emptying How often have you had the sensation of not emptying your bladder? 0 1 2 3 4 5
  2. Frequency How often have you had to urinate less than every two hours? 0 1 2 3 4 5
  3. Intermittency How often have you found you stopped and started again several times when you urinated? 0 1 2 3 4 5
  4. Urgency How often have you found it difficult to postpone urination? 0 1 2 3 4 5
  5. Weak Stream How often have you had a weak urinary stream? 0 1 2 3 4 5
  6. Straining How often have you had to strain to start urination? 0 1 2 3 4 5 None 1 Time 2 Times 3 Times 4 Times 5 Times
  7. Nocturia How many times did you typically get up at night to urinate? 0 1 2 3 4 5
post voiding residual urine | 1 year
  Post-void residual urine (PVR) is the amount of urine that remains in the bladder after urinating. It can be estimated by ultrasound or measured by catheterization1. A small amount of PVR is normal, but a high amount can indicate a urinary obstruction or other problems

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elshazly M, Sultan S, Shaban M, Zanaty F. Evaluation of a novel technique of bladder neck and supramontanal sparing ejaculatory preserving transurethral prostatectomy. World J Urol. 2021 Nov;39(11):4215-4219. doi: 10.1007/s00345-021-03752-z. Epub 2021 Jun 6. PMID 34091741
- [Background] Brant A, Cho A, Posada Calderon L, Te A, Kashanian J, Chughtai B. Ejaculatory Hood-Sparing Vaporization of the Prostate and Its Impact on Erectile, Ejaculatory, and Sexual Function. Urology. 2020 Oct;144:177-181. doi: 10.1016/j.urology.2020.06.072. Epub 2020 Jul 23. PMID 32711008